CLINICAL TRIAL: NCT02653443
Title: A Randomized, Multi-center, Open-label, Paired Controlled, Crossover In Vivo Study to Assess the Recovery and Lifespan of Radiolabeled Autologous INTERCEPT Treated Apheresis Platelet Components Suspended in Nominal 35% Plasma and 65% InterSol Stored for 6 or 7 Days
Brief Title: A Randomized, Multi-center, Open-label, Paired Controlled, Crossover In Vivo Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLI 00116
Record Dates: First submitted 2015-12-02; First posted 2016-01-12 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: INTERCEPT; Platelet; Pathogen Inactivation; Platelets Components Stored; Therapeutic Efficacy
MeSH Terms: interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 6 (Experimental): Each subject will provide two apheresis platelet donations (one per period) and receive two infusions (one per period) of autologous radiolabeled fresh platelets combined with INTERCEPT treated platelet components stored for either 6 or 7 days (approximately 10 to 30 mL).
  Interventions: Biological: Autologous apheresis Platelet Components, prepared with the INTERCEPT Blood System for Platelets.; Biological: Autologous apheresis Conventional untreated Platelet Components
- Day 7 (Experimental): Each subject will provide two apheresis platelet donations (one per period) and receive two infusions (one per period) of autologous radiolabeled fresh platelets combined with conventional untreated platelet components stored for either 6 or 7 days (approximately 10 to 30 mL).
  Interventions: Biological: Autologous apheresis Platelet Components, prepared with the INTERCEPT Blood System for Platelets.; Biological: Autologous apheresis Conventional untreated Platelet Components

INTERVENTIONS:
Biological: Autologous apheresis Platelet Components, prepared with the INTERCEPT Blood System for Platelets. — Each subject will provide two apheresis platelet donations (one per period) and receive two infusions (one per period) of autologous radiolabeled fresh platelets combined with INTERCEPT treated platelet components stored for either 6 or 7 days (approximately 10 to 30 mL). Platelets are administered by intravenous infusion in a peripheral vein via 19-gauge butterfly infusion needle.
Biological: Autologous apheresis Conventional untreated Platelet Components — Each subject will provide two apheresis platelet donations (one per period) and receive two infusions (one per period) of autologous radiolabeled fresh platelets combined with conventional untreated platelet components stored for either 6 or 7 days (approximately 10 to 30 mL). Platelets are administered by intravenous infusion in a peripheral vein via 19-gauge butterfly infusion needle.

SUMMARY:
The objective of this study is to test the hypothesis that INTERCEPT Blood System for platelet components stored for 6 or 7 days after INTERCEPT Blood System treatment retain sufficient viability for therapeutic efficacy. The post-infusion recovery and lifespan of autologous INTERCEPT Blood System for platelet components in 35% plasma/65% InterSol (Test platelets) stored for 6 or 7 days will be measured in comparison to "fresh" autologous radiolabeled platelets (Control platelets) according to FDA guidance for platelet testing (FDA 1999). Recovery and lifespan results between components stored for 6 and 7 days will also be assessed.

DETAILED DESCRIPTION:
For each of the 2 study donation periods, this study will have the following procedures: single or double dose platelet apheresis collection, pathogen inactivation with INTERCEPT Blood System treatment, storage for 6 or 7 days (depending on the period and randomization scheme) at 20°C to 24°C with agitation, collection of "fresh" autologous platelets, radiolabeling, infusion of fresh and stored INTERCEPT Blood System-treated radiolabeled autologous platelets, and collection of blood samples for assessment of platelet recovery and survival (lifespan). There will be a minimum wash-out period of two weeks between the two study periods.

Apheresis platelets will be collected using the Amicus separator and stored for 6 or 7 days (depending on the period and randomization scheme) in 35% plasma/65% InterSol.

Procedures will be as follows: On Day 0, each healthy volunteer subject has apheresis platelets collected. INTERCEPT Blood System treatment will begin on either the day of donation (Day 0) or the day following donation (Day 1) and will be completed within 24 hours after collection. Platelets will then be stored for 6 or 7 days after collection (depending on the period and randomization scheme) at 22°C ±2°C with agitation. Aliquots for in vitro platelet function will be taken on Day 0/1 before INTERCEPT Blood System treatment and on Day 6 or 7. On Day 6 or 7, healthy volunteers will return to the site, and 43 mL of blood will be drawn into a syringe containing 9 mL of Anticoagulant Citrate Dextrose Solution, Formula A (ACD-A). Fresh platelets will be prepared from this sample. An aliquot (10-20 mL) of the stored INTERCEPT Blood System for platelets will be aseptically removed from each subject's test container.

Previously stored (Test) and fresh (Control) platelets will be radiolabeled according to randomization assignment with either Chromium-51 (51Cr) (≤20 μCi) as sodium radiochromate (Na251CrO4) or Indium-111 (111In) (≤15 μCi) as indium oxine, following the labeling and washing procedures outlined by the Biomedical Excellence for Safer Transfusion (BEST) Collaborative. The isotope labels will be assigned randomly with equal probability that fresh platelets and stored INTERCEPT Blood System for platelets will be labeled with each isotope., and the same randomization assignment of isotope labels will be utilized for both donation periods for the same subject. Aliquots of the fresh and stored platelets will be radiolabeled in tubes with the standard techniques. After radiolabeling, the autologous fresh and stored INTERCEPT Blood System for platelets will be simultaneously infused into the subject (approximately 10-30 mL). Negative pregnancy test for females of childbearing potential are required before infusion.

Blood samples for radioactivity measurements will be drawn immediately before infusion and at approximately 0, 0.5, 1, and 2 hours post-infusion, and then 6 more samples will be drawn at 1, 2, 3, 4 (or 6), 7, and 11±1 days post-infusion, at approximately the same time of day as the radiolabeled platelet infusion was administered (±4 hours).

Patients will be monitored for safety (adverse events) from the beginning of the study until 10 days following the infusion of radiolabelled platelets in period 2.

Radioactivity measurements Samples will be obtained from the radiolabeled fresh and stored INTERCEPT Blood System for platelets before infusion and used as a radioactive standard. By measuring the volume infused, the total dose of radioactivity infused will be calculated. In vitro elution of the label from the transfused platelets will be determined by the BEST elution assessment method, as well as the in vivo elution of radioactivity from the serial blood samples obtained post-infusion of the labeled platelets.

The standard as well as the subject's whole-blood samples will be corrected for elution and also for the residual activity in the cellular fraction one day after the infusion. Data points 24 hours post-infusion will be used to calculate in vivo recovery after all radioactive corrections have been made. The radioactivity of the samples will be determined by use of a gamma counter. A multiple-hit model will be used to estimate the survival of the radioactively labeled platelets.

ELIGIBILITY:
Inclusion Criteria:

* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam)
* Meet FDA, American Association of Blood Banks (AABB), and site guidelines for blood donation or apheresis platelet donation
* Complete blood count (CBC) and serum chemistry values within established reference ranges or within guidelines as above.
* Pre-donation platelet count of more than 150×10^9 platelets/L
* Negative blood donor screening test panel for Human Immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human T-Lymphotropic virus (HTLV), syphilis, and West Nile virus (WNV)
* Male and female subjects of childbearing potential must agree to use a medically acceptable method of contraception throughout the study. A barrier method of contraception must be included, regardless of other methods.
* Signed and dated informed consent form

Exclusion Criteria:

* Clinically significant acute or chronic disease (as determined by the Investigator)
* Pregnant or nursing females
* Male or female subjects of childbearing potential not using effective contraception
* Disease states or conditions that preclude blood donation or apheresis platelet donation per AABB reference standards
* Treatment with aspirin or aspirin-containing medications within 7 days of apheresis or treatment with non-steroidal anti inflammatory drugs (NSAID), anti-platelet agents or other drugs affecting platelet viability within 3 days of apheresis (e.g. ibuprofen or other NSAIDs)
* Subject received platelet inhibitor within 14 days of donation (e.g. clopidogrel, ticlopidine)
* Splenectomized subjects
* History of known hypersensitivity to indium or chromium
* Participation in another clinical study currently or within the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Post infusion recovery of the Test platelets compared to fresh platelets. | 16 Days
Post infusion recovery of the Test platelets compared to fresh platelets. | 17 Days
Post infusion lifespan of Test platelets compared to fresh platelets. | 16 Days
Post infusion lifespan of Test platelets compared to fresh platelets. | 17 Days
Adverse events: any untold medical occurrence in a subject or clinical investigation subject administered an investigational product and which does not necessarily have a causal relationship with this treatment. | 16 Days
Adverse events: any untold medical occurrence in a subject or clinical investigation subject administered an investigational product and which does not necessarily have a causal relationship with this treatment. | 17 Days
Body Mass Index (kg/m^2) | 16 Days
Body Mass Index (kg/m^2) | 17 Days
Hematocrit (g/dL) | 16 Days
Hematocrit (g/dL) | 17 Days
Hemoglobin (g/dL) | 16 Days
Hemoglobin (g/dL) | 17 Days
Red Blood Cell Count (x10^12/L) | 16 Days
Red Blood Cell Count (x10^12/L) | 17 Days
Platelet Count (×10^3μL) | 16 Days
Platelet Count (×10^3μL) | 17 Days
White Blood Cell Count - with Differential (x10^9/L) | 16 Days
White Blood Cell Count - with Differential (x10^9/L) | 17 Days
Blood Urea Nitrogen (mg/dL) | 16 Days
Blood Urea Nitrogen (mg/dL) | 17 Days
Calcium (mg/dL) | 16 Days
Calcium (mg/dL) | 17 Days
Chloride (mEq/L) | 16 Days
Chloride (mEq/L) | 17 Days
Creatinine (mg/dL) | 16 Days
Creatinine (mg/dL) | 17 Days
Glucose (mg/dL) | 16 Days
Glucose (mg/dL) | 17 Days
Potassium (mEq/L) | 16 Days
Potassium (mEq/L) | 17 Days
Sodium (mEq/L) | 16 Days
Sodium (mEq/L) | 17 Days
Post infusion recovery of the platelets at Day 6 platelets compared to Day 7 platelets. | 16 Days
Post infusion recovery of the platelets at Day 6 platelets compared to Day 7 platelets. | 17 Days
Post infusion lifespan of the platelets at Day 6 platelets compared to Day 7 platelets. | 16 Days
Post infusion lifespan of the platelets at Day 6 platelets compared to Day 7 platelets. | 17 Days

SECONDARY OUTCOMES:
pH (pH) | 16 Days
pH (pH) | 17 Days
Platelet count (×10^3/μL) | 16 Days
Platelet count (×10^3/μL) | 17 Days
Platelet dose (×10^11 cells/component) | 16 Days
Platelet dose (×10^11 cells/component) | 17 Days
Mean platelet volume (MPV) (fL) | 16 Days
Mean platelet volume (MPV) (fL) | 17 Days
Morphology score (Kunicki Score) | 16 Days
Morphology score (Kunicki Score) | 17 Days
Component volume (mL) | 16 Days
Component volume (mL) | 17 Days
Glucose (mmol/L) | 16 Days
Glucose (mmol/L) | 17 Days
Lactate (mmol/L) | 16 Days
Lactate (mmol/L) | 17 Days
pO2 (mm Hg) | 16 Days
pO2 (mm Hg) | 17 Days
pCO2 (mm Hg) | 16 Days
pCO2 (mm Hg) | 17 Days
Bicarbonate (HCO3-) (mmol/L) | 16 Days
Bicarbonate (HCO3-) (mmol/L) | 17 Days
Lactate dehydrogenase (IU/L) | 16 Days
Lactate dehydrogenase (IU/L) | 17 Days
Hypotonic Shock Response (HSR) (%) | 16 Days
Hypotonic Shock Response (HSR) (%) | 17 Days
Extent of Shape Change (ESC) (%) | 16 Days
Extent of Shape Change (ESC) (%) | 17 Days
p-selectin expression (CD62) (% activation) | 16 Days
p-selectin expression (CD62) (% activation) | 17 Days
Adenosine 5'-Triphosphate (ATP) (nmol/10^8 platelets) | 16 Days
Adenosine 5'-Triphosphate (ATP) (nmol/10^8 platelets) | 17 Days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hoxworth Blood Center, Cincinnati, Ohio